CLINICAL TRIAL: NCT04818086
Title: Phase Ib/2a Drug-drug Interaction Study of Lemborexant as an Adjunctive Treatment for Buprenorphine/Naloxone for Opioid Use Disorder
Brief Title: Drug-drug Interaction Study of Lemborexant as an Adjunctive Treatment for Buprenorphine/Naloxone for Opioid Use Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20021136; UG1DA050207 (NIH)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Drug Interaction; Analgesics; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lemborexant; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lemborexant Arm (Active Comparator): Study Drug Dosage: 5 mg of lemborexant (Time 1) , and 10 mg of lemborexant (Time 2) combined with 16 mg/4 mg of buprenorphine-naloxone sublingually as a film.
  Interventions: Drug: Lemborexant; Drug: Buprenorphine-naloxone
- Placebo Arm (Placebo Comparator): Comparative placebo combined with 16 mg/4 mg of buprenorphine-naloxone sublingually as a film (at both Time 1 and Time 2)
  Interventions: Drug: Placebo; Drug: Buprenorphine-naloxone

INTERVENTIONS:
Drug: Lemborexant — Participants will complete 2 inpatient visits which may last up to 24 hours. The two visits will be approximately 14 days apart. During the inpatient visit they will receive 5 mg of lemborexant (first visit) and 10 mg of lemborexant (second visit).
  Other Names: Dayvigo
  Arms: Lemborexant Arm
Drug: Placebo — Participants will complete 2 inpatient visits which may last up to 24 hours. The two visits will be approximately 14 days apart. During the inpatient visit they will receive a placebo which is encapsulated to look the same as the intervention drug.
  Arms: Placebo Arm
Drug: Buprenorphine-naloxone — Participants will receive 16 mg/4 mg of buprenorphine-naloxone sublingually as a film.

SUMMARY:
The purpose of this research study is to test the safety, tolerability, drug interactions with buprenorphine-naloxone, and effectiveness lemborexant when used to treat Opioid Use Disorder.

DETAILED DESCRIPTION:
The purpose of this study is to test the effects of lemborexant when used in combination with opioids (including buprenorphine). We are also interested in learning lemborexant might help improve sleep problems and problems related to opioid use (e.g., cravings, withdrawal), in people with opioid use disorder. Study participants will be randomly assigned in a two to one ratio to receive either lemborexant or placebo. Lemborexant (DAYVIGO®) is approved by the U. S. Food and Drug Administration (FDA) for treatment of insomnia.

In this study, Participants will be asked to do the following things:

1. Visit the CARI clinic and/or Motivate clinic at Jackson Center to complete study screening.
2. Visit the VCUHS Clinical Research Unit to complete an outpatient blood draw/testing visit.
3. Take either lemborexant or the placebo, depending upon which group subjects are assigned to.
4. Complete two (2) overnight study visits at the VCUHS Clinical Research Unit.
5. Complete 8 outpatient follow-up visits (broken into 2 four day visit groupings)
6. Have an EKG during screening and at each study visit (outpatient and inpatient)
7. Have an IV inserted into your arm for blood draws at the outpatient blood draw visit and each inpatient visit.
8. Record sleep in a sleep diary.
9. Take surveys and answer questions about health, mental health, medications used, drug use, and cravings.
10. Complete tasks on the computer.
11. Complete physical exams during screening, outpatient and inpatient visits.
12. Give permission for the researchers to collect information about opioid treatment, medical status, and other information from your medical record.

Participation in this study will last approximately 4 weeks. Approximately 18 people will participate in the drug interaction phase of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 - 65 years-of-age;
2. Understand the study procedures and provide written informed consent in English language;
3. Meet current DSM-5 criteria for opioid use disorder, of at least moderate severity, currently engaged medication assisted treatment at a buprenorphine-naloxone sublingual film daily dose ranging from 8mg/2mg to 24mg/6mg or buprenorphine sublingual tablet 5.7mg/1.4mg to 17.1/4.3 once daily for at least last 2 weeks;
4. Have a positive urine drug screen for buprenorphine during screening and on admission to the clinical research unit to document buprenorphine use;
5. Have a Pittsburgh Sleep Quality Index (PSQI) Total Score of 6 or higher.

Exclusion Criteria:

1. Contraindications for participation as determined by medical history and physical exam performed by study NP or study physician;
2. Pregnant or nursing women;
3. Baseline ECG with clinically significant abnormal conduction;
4. Uncontrolled serious psychiatric or major medical disorder, including COPD. Narcolepsy is also considered exclusionary;
5. Taking prescription or over-the counter drugs or dietary supplements known to significantly inhibit CYP3A4 (such as Clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir), or CYP3A4 inducers (such as phenobarbital, phenytoin, rifampicin, St. John's Wort, and glucocorticoids);
6. Prescribed medications for insomnia, or unable to discontinue over the counter drugs or dietary supplements used to treat insomnia on study days.
7. Current severe alcohol use disorder or current benzodiazepine use disorder
8. Current DSM-5 diagnosis of any psychoactive substance use disorder other than opioids, cocaine, marijuana, or nicotine, or mild or moderate alcohol use disorder. Diagnosis of mild to moderate use disorder for alcohol will not be considered exclusionary.
9. Any previous medically adverse reaction to opioids or lemborexant:
10. Significant current suicidal or homicidal ideation (C-SSRS "yes" answers on questions 4 or 5) or a history of suicide attempt within the past 6 months.
11. Subjects with Suicidal Behaviors Questionnaire-Revised score ≥8 at the screening visit.
12. Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Comparative placebo combined with 16 mg/4 mg of buprenorphine-naloxone sublingually as a film (at both Time 1 and Time 2)
  Placebo: Participants will complete 2 inpatient visits which may last up to 24 hours. The two visits will be approximately 14 days apart. During the inpatient visit they will receive a placebo which matches the intervention drug.
  Buprenorphine-naloxone: Participants will receive 16 mg/4 mg of buprenorphine-naloxone sublingually as a film.
Period: Overall Study
Arm/Group | Lemborexant Arm | Placebo Arm
Started | 12 | 6
Completed | 11 | 5
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lemborexant Arm | Placebo Arm | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (7.3) | 44.3 (14) | 39.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 6 | 17
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 9 | 2 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulse Oximetry During the Baseline Visit
Description: A finger pulse oximeter will be used to assess oxygen saturation (%). Change is calculated from the pulse oximetry readings from pre to post medication/placebo dose administered during the baseline study visit, this is a safety measure.
Time Frame: Baseline visit (Safety measure)
Population: Baseline
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
percentage of oxygen saturation | -0.17 (.94) | -0.33 (.82)

2. Primary Outcome: Change in Pulse Oximetry During Week 1 Visit
Description: A finger pulse oximeter will be used to asses pulse oximetry. Change is calculated from the pulse oximetry readings from pre to post medication/placebo dose administered during the study visit (safety measure)
Time Frame: Week 1 visit, safety measure
Population: Week 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
percentage of oxygen saturation | -0.17 (1.94) | -0.50 (1.05)

3. Primary Outcome: Change in Pulse Oximetry During Week 2 Visit
Description: A finger pulse oximeter will be used to assess pulse oximetry. Change is calculated from the pulse oximetry readings from pre to post medication/placebo dose administered during the study visit. This is a safety measure.
Time Frame: Week 2 visit, safety measure
Population: Week 2
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
percentage of oxygen saturation | -0.27 (1.49) | -0.20 (0.84)

4. Primary Outcome: Change in Blood Pressure During Baseline Study Visit
Description: Blood Pressure measured with an automatic BP cuff. Change is calculated from the blood pressure readings from pre to post medication/placebo dose administered during the study visit. This is a safety measure.
Time Frame: Baseline Visit, safety measure
Population: Baseline
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
mmHg (millimeters of mercury) | -9.42 (10.40) | -2.50 (12.29)

5. Primary Outcome: Change in Blood Pressure During Week 1 Study Visit
Description: as for outcome 4
Time Frame: Week 1 visit, safety measure
Population: Week 1
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
mmHg (millimeters of mercury) | -6.58 (6.64) | -4.50 (5.68)

6. Primary Outcome: Change in Blood Pressure During Week 2 Study Visit
Description: as for outcome 4
Time Frame: Week 2 visit, safety measure
Population: Week 2
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
mmHg (millimeters of mercury) | 1.09 (12.85) | -3.60 (8.53)

7. Primary Outcome: Change in Patient Consciousness During the Baseline Visit
Description: The Richmond Agitation Sedation Scale (RASS) measures level of patient consciousness on a 10 point scale ranging from plus +4 (combative/agitated) to minus 5 (unarousable/sedated). Change is calculated from the RASS assessment scores obtained from pre to post medication/placebo dose administered during the study visit. This is a safety measure. RASS is one of the most commonly used scales to determine the sedation level, and it measures the severity of agitation and sedation with a score of +4 to -5: +4: combative, +3: very agitated, +2: agitated, +1: restless, 0: alert and calm, -1: drowsy, -2: light sedation, -3: moderate sedation, -4: deep sedation, and -5 unarousable. A positive score is preferable to a negative score.
Time Frame: Baseline visit, safety measure
Population: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -0.17 (0.39) | 0 (.63)

8. Primary Outcome: Change in Patient Consciousness During the Week 1 Study Visit
Description: The Richmond Agitation Sedation Scale (RASS) measures level of patient consciousness on a 10 point scale ranging from plus 4 (combative/agitated) to minus 5 (unarousable/sedated).Change is calculated from the RASS assessment scores obtained from pre to post medication/placebo dose administered during the study visit. This is a safety measure. RASS is one of the most commonly used scales to determine the sedation level, and it measures the severity of agitation and sedation with a score of +4 to -5: +4: combative, +3: very agitated, +2: agitated, +1: restless, 0: alert and calm, -1: drowsy, -2: light sedation, -3: moderate sedation, -4: deep sedation, and -5 unarousable. A positive score is preferable to a negative score.
Time Frame: Week 1 visit, safety measure
Population: week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | 0.00 (0.60) | 0.33 (0.52)

9. Primary Outcome: Change in Patient Consciousness
Description: The Richmond Agitation Sedation Scale (RASS) measures level of patient consciousness on a 10 point scale ranging from plus 4 (combative/agitated) to minus 5 (unarousable/sedated). Change is calculated from the RASS assessment scores obtained from pre to post medication/placebo dose administered during the study visit. This is a safety measure. RASS is one of the most commonly used scales to determine the sedation level, and it measures the severity of agitation and sedation with a score of +4 to -5: +4: combative, +3: very agitated, +2: agitated, +1: restless, 0: alert and calm, -1: drowsy, -2: light sedation, -3: moderate sedation, -4: deep sedation, and -5 unarousable. A positive score is preferable to a negative score.
Time Frame: Week 2 visit, safety measure
Population: week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
score on a scale | -0.18 (0.87) | -0.20 (0.45)

10. Primary Outcome: Change in Buprenorphine Plasma Concentration (PK) During the Baseline Visit
Description: Blood will be drawn pre-dose and at specific time points (8, 8:30, 10, 12 and 4pm) to determine the area under the plasma concentration-time curve for buprenorphine.
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 0
Nanograms/milliliter (ng/mL) | 0.26 (0.29) |

11. Primary Outcome: Change in Buprenorphine Plasma Concentration (PK) During Week 1 Study Visit
Description: as for outcome 10
Time Frame: Week 1
Population: Week 1
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 0
Nanograms/milliliter (ng/mL) | 0.15 (0.18) |

12. Primary Outcome: Change in Buprenorphine Plasma Concentration (PK) During Week 2 Study Visit
Description: as for outcome 10
Time Frame: Week 2
Population: Week 2
Measure: Mean (Standard Deviation); unit: Nanograms/milliliter (ng/mL)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 0
Nanograms/milliliter (ng/mL) | 0.12 (0.18) |

13. Primary Outcome: Change in Lemborexant PK During Baseline Study Visit
Description: Blood will be drawn pre-dose and at specific time points (8, 8:30, 10, 12 and 4pm) to determine the peak plasma concentration for Lemborexant.
  Currently, we have no pathway to obtain the lorcaserin PK results. The reason for that is the methods used for the original lorcaserin human PK testing are proprietary and we would have to re-do all of that research ourselves, which is outside the scope of what we are able to do.
Time Frame: Baseline visit
Population: Lemborexant serum levels are not provided as the detailed methods for lemborexant level determination are proprietary and we do not have access to those methods. Hence, we are not able to provide the lemborexant levels. Currently, we have no pathway to obtain the lorcaserin PK results. The reason for that is the methods used for the original lorcaserin human PK testing are proprietary and we would have to re-do all of that research ourselves, which is outside the scope of what we are able to do.
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Change in Lemborexant PK During Week 1 Study Visit
Description: Blood will be drawn pre-dose and at specific time points (8, 8:30, 10, 12 and 4pm) to determine the area under the plasma concentration-time curve for Lemborexant. Currently, we have no pathway to obtain the lorcaserin PK results. The reason for that is the methods used for the original lorcaserin human PK testing are proprietary and we would have to re-do all of that research ourselves, which is outside the scope of what we are able to do.
Time Frame: Week 1 visit
Population: as for outcome 13
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Change in Lemborexant PK During Week 2 Study Visit
Description: as for outcome 13
Time Frame: Week 2 visit
Population: as for outcome 13
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change in Respiration During the Baseline Study Visit (Pre- to Post-dose)
Description: Respiration will be measured with End Title CO2( EtC02) which is a measure of CO2 (measured in millimeters of mercury, "mmHg") plotted against time. Participants will wear a mask which will be connected to a Capnographer. End Title CO2 should be between 35-45 mmHg with box wave form.
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
mmHg (millimeters of mercury) | 1.0 (4.18) | 1.40 (3.65)

17. Primary Outcome: Change in Respiration During the Week 1 Study Visit (Pre- to Post-dose)
Description: as for outcome 16
Time Frame: Week 1 visit
Population: Week 1
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
millimeters of mercury (mmHg) | 1.67 (2.46) | 0.50 (8.80)

18. Primary Outcome: Change in Respiration During Week 2 Study Visit (From Pre- to Post-dose)
Description: as for outcome 16
Time Frame: Week 2 visit
Population: Week 2
Measure: Mean (Standard Deviation); unit: mmHg (millimeters of mercury)
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
mmHg (millimeters of mercury) | 2.18 (3.28) | 1.60 (1.52)

19. Secondary Outcome: Change in Drug Effects During Baseline Study Visit (Pre- to Post- Dose)
Description: Drug effects will be assessed using the Drug Effects Questionnaire (DEQ). The DEQ is comprised of 11 items which assess physical effects of the drug. Participants rate each physical effect on a visual analog scale from "not at all" (0) to "extremely" (100). A higher score indicates greater drug effect. The Drug Effects Questionnaire (DEQ) is widely used in studies of acute subjective response (SR) to a variety of substances and assesses the extent to which participants (1) feel any substance effect(s), (2) feel high, (3) like the effects, (4) dislike the effects, and (5) want more of the substance using 100mm Visual Analog Scales.
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | 21.0 (39.95) | 7.33 (8.91)

20. Secondary Outcome: Change in Drug Effects During Week 1 Study Visit (Pre- to Post- Dose)
Description: as for outcome 19
Time Frame: Week 1 visit
Population: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | 14.50 (21.72) | 5.33 (35.83)

21. Secondary Outcome: Change in Drug Effects During Week 2 Study Visit (Pre- to Post Dose)
Description: as for outcome 19
Time Frame: Week 2 visit
Population: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
score on a scale | 5.45 (41.31) | 18.00 (32.27)

22. Secondary Outcome: Change in Opioid Craving During Each Visit (Pre- to Post- Dose)
Description: Opioid craving will be measured by a Brief Substance craving scale (BSCS). The BSCS is a 16 item, self-report instrument assesses craving for substances of abuse over a 24 hour period. Intensity and frequency of craving are recorded on a five-point Likert scale, with higher scores indicating greater craving. 0-none at all, 1- slight, 2-moderate, 3-considerable, 4-extreme.
Time Frame: During each inpatient visit (baseline through week 2) from admission to discharge at each visit, up to 24 hours
Population: During each inpatient visit from admission to discharge, up to 24 hours (Baseline through week 2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -025 (2.09) | 3.0 (8.0)

23. Secondary Outcome: Change in Opioid Withdrawal Effects During Baseline Visit (Pre- to Post- Dose)
Description: Opioid withdrawal symptoms will be measured with the Subjective Opioid Withdrawal Scale (SOWS). The SOWS contains 16 likert scaled items with participant rate from 0 (not at all), 1(slight), 2 (moderate), 3 (considerable) to 4 (Extreme). A higher score indicates higher opioid withdrawal effects (Range 0-64).
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -1.92 (2.39) | -.033 (0.52)

24. Secondary Outcome: Change in Opioid Withdrawal Effects During Week 1 Visit (Pre- to Post- Dose)
Description: Opioid withdrawal symptoms will be measured with the Subjective Opioid Withdrawal Scale (SOWS). The SOWS contains 16 likert scaled items with participant rate from 0 (not at all), 1(slight), 2 (moderate), 3 (considerable) to 4 (Extremely). A higher score indicates higher opioid withdrawal effects(Range 0-64).
Time Frame: Week 1 visit
Population: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -0.25 (0.97) | -0.17 (0.41)

25. Secondary Outcome: Change in Opioid Withdrawal Effects During Week 2 Visit (Pre- to Post- Dose)
Description: Opioid withdrawal symptoms will be measured with the Subjective Opioid Withdrawal Scale (SOWS). The SOWS contains 16 likert scaled items with participant rate from 0 (not at all), 1(slight), 2 (moderate), 3 (considerable) to 4 (Extremely). A higher score indicates higher opioid withdrawal effects (Range 0-64).
Time Frame: Week 2 visit
Population: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
score on a scale | -0.45 (0.93) | 0 (0)

26. Secondary Outcome: Change in Objective Opioid Withdrawal During Baseline Study Visit (Pre- to Post- Dose)
Description: Participants will be assessed by research staff using the Clinical Opioid Withdrawal Scale (COWS) which consists of 11 items. A higher score indicates greater withdrawal effects. (COWS, range 0-48). 5-12=mild, 13-24=moderate, 25-36=moderate severe, and more than 36=severe withdrawal.
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -0.83 (1.19) | -0.17 (0.98)

27. Secondary Outcome: Change in Objective Opioid Withdrawal During Week 1 Study Visit (Pre- to Post-dose)
Description: Participants will be assessed by research staff using the Clinical Opioid Withdrawal Scale (COWS) which consists of 11 items. A higher score indicates greater withdrawal effects(COWS, range 0-48). 5-12=mild, 13-24=moderate, 25-36=moderate severe, and more than 36=severe withdrawal.
Time Frame: Week 1 visit
Population: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | -0.50 (1.09) | -0.17 (0.41)

28. Secondary Outcome: Change in Objective Opioid Withdrawal During Week 2 Study Visit (Pre- to Post- Dose)
Description: Participants will be assessed by research staff using the Clinical Opioid Withdrawal Scale (COWS) which consists of 11 items. A higher score indicates greater withdrawal effects (COWS, range 0-48). 5-12=mild, 13-24=moderate, 25-36=moderate severe, and more than 36=severe withdrawal.
Time Frame: Week 2 visit
Population: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
score on a scale | -0.27 (1.27) | 0 (0)

29. Secondary Outcome: Impulsivity
Description: Impulsivity is measured by a delayed discounting task (DDT). Participants are presented with a series of choices and will choose to receive pretend money now or after a delay. The task yields a discounting rate. Higher discounting rates indicate greater impulsivity. Delay discounting, the tendency to choose small, immediate rewards over larger, delayed rewards is robustly associated with substance use. The longer the timeframe that the subject delays the rewards, the larger the reward.
Time Frame: Baseline visit
Population: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | 55.73 (90.25) | 74.74 (51.31)

30. Secondary Outcome: Impulsivity
Description: as for outcome 29
Time Frame: Week 1 visit
Population: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 12 | 6
score on a scale | 6.51 (76.73) | 22.92 (23.96)

31. Secondary Outcome: Impulsivity
Description: as for outcome 29
Time Frame: Week 2 visit
Population: Week 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lemborexant Arm | Placebo Arm
Number analyzed (Participants) | 11 | 5
score on a scale | -40.63 (126.27) | -1.25 (9.47)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the second week scheduled visit.
Arm/Group | Lemborexant Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 6/12 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lemborexant Arm (N=12) | Placebo Arm (N=6)
Assaulted (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tongue numbness (Nervous system disorders) | 0 (0) | 1 (1)
Nausea/vomiting/diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
sleep paralysis (Nervous system disorders) | 1 (1) | 0 (0)
back/shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
skin/soft tissue irriatation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
arthritis flare (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04818086/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04818086/ICF_001.pdf